CLINICAL TRIAL: NCT04508205
Title: Effectiveness of CGB-400 (Cosmetic) for the Reduction of Facial Redness and Bumps and Blemishes
Brief Title: CGB-400 for the Reduction of Facial Redness and Bumps and Blemishes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CAGE Bio Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGB-400-001a
Record Dates: First submitted 2020-08-02; First posted 2020-08-11 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with redness and bumps and/or blemishes (Experimental): Topical administration twice daily for 12 weeks
  Interventions: Drug: CGB-400

INTERVENTIONS:
Drug: CGB-400 — BID application

SUMMARY:
Open-label multicenter study using CGB-400 Gel to reduce facial redness, bumps, and blemishes.

DETAILED DESCRIPTION:
This is a Open-label multicenter study to evaluate the ability of CGB-400 Gel to reduce facial redness and bumps/blemishes typically associated with rosacea. Approximately 25 subjects will be enrolled.

Subjects will receive study treatment for 12 weeks and attend a total of 5 study visits (i.e., BL, W2, W4, W8, W12).

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient, male or female of any race, 18 years of age or older. Female subjects of childbearing potential must have a negative UPT at Baseline and practice a reliable method of contraception throughout the study.
2. Facial redness associated with rosacea with or without bumps or blemishes.
3. Facial redness (IGA-R) score of 2 or 3 (i.e., mild or moderate).
4. IGA score of 2 or 3 (i.e., mild or moderate).
5. Absence of any skin conditions that could interfere with the visual erythema assessments.
6. Willing to forego any other topical or non-topical treatment on the study areas during treatment (other than sun protection or the study specified face wash and moisturizer).
7. Willing to use the provided skincare regimen (e.g., face wash and moisturizer) over the duration of the study.
8. Sign the IRB-approved ICF (which includes HIPAA) prior to any study-related procedures being performed.

Exclusion Criteria:

1. Known hypersensitivity or previous allergic reaction to any constituent of the Investigational Products (i.e., essential oils, fragrance, choline, phosphatidylcholine, etc.).
2. Any transient flushing syndrome.
3. History of basal cell carcinoma within 6 months of Visit 1.
4. History or presence of a skin condition/disease that is located in the treatment area(s) and might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, psoriasis, significant actinic damage, vitiligo, open wounds, infection, etc.).
5. Diagnosis of severe rosacea, ocular rosacea, rhinophymatous rosacea, or acne fulminans at Baseline.
6. Blepharitis/meibomianitis requiring systemic treatment by an ophthalmologist.
7. Uncontrolled systemic disease.
8. Foreseen unprotected and intense/excessive UV exposure during the course of the study.
9. Use of any of the following concomitant medications/procedures:

   * Cosmetic and/or OTC products for redness reduction and/or skin clearing
   * Topical medications for rosacea
   * Systemic antibiotics or corticosteroids
   * Topical antibiotics, corticosteroids, or antiparasitic agents
   * Intense/excessive ultraviolet (UV) radiation
   * Phototherapy, energy-based therapy, facials, chemical peels, microdermabrasion
10. Exposure to any other investigational drug/device within 30 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment (IGA) | Week 12
  5-point scale (0 - Clear skin with no signs of bumps/blemishes; 1 - Almost clear; minimal lesions (<5 bumps/blemishes); 2 - Mild facial lesions (6-10 bumps/blemishes): 3 - Moderate lesions; marked redness (11-25 bumps/blemishes): 4 - Severe lesions; fiery redness (>25 bumps/blemishes)
Investigator's Global Assessment of Redness (IGA-R) | Week 12
  5-point scale (0 - Clear skin with no signs of redness to 4 - Severe; fiery redness)

SECONDARY OUTCOMES:
Investigator's Global Assessment (IGA) | Day 0, Week 2, Week 4, Week 8
  5-point scale (0 - Clear skin with no signs of bumps/blemishes; 1 - Almost clear; minimal lesions (<5 bumps/blemishes); 2 - Mild facial lesions (6-10 bumps/blemishes): 3 - Moderate lesions; marked redness (11-25 bumps/blemishes): 4 - Severe lesions; fiery redness (>25 bumps/blemishes)
Investigator's Global Assessment of Redness (IGA-R) | Day 0, Week 2, Week 4, Week 8
  5-point scale (0: no redness; 1: slight redness; 2: Definite redness; 3: Marked redness and 4: Fiery redness)
Bumps/Blemishes Count | Day 0, Week 2, Week 4, Week 8, Week 12
  Numerical count of Bumps/Blemishes
Patient Global Assessment | Day 0, Week 2, Week 4, Week 8, Week 12
  5-point scale (0: excellent effectiveness; 1: good effectiveness; 2: Effective; 3: No significant benefit and 4: No benefit at all)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cage Bio Investigative Site 1, Fremont, California
  - Cage Bio Investigative Site 2, San Diego, California
  - Cage Bio Investigative Site 3, Edgewater, Florida

IPD SHARING:
Plan to Share IPD: No